CLINICAL TRIAL: NCT03854500
Title: A Randomised Trial of Tenecteplase vs. Alteplase in Acute Ischemic Stroke
Brief Title: The Norwegian Tenecteplase Stroke Trial 2
Acronym: NOR-TEST 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per protocol safety analysis 200 patients showed a significant difference in bleeding rates between the two drug groups.
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-003090-95
Record Dates: First submitted 2019-01-21; First posted 2019-02-26 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Acute; Cerebrovascular Disorders; Ischemic Stroke
Keywords: Tenecteplase; Thrombolysis; Alteplase
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Ischemic Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: Randomized, controlled multicenter study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenecteplase (Active Comparator): Tenecteplase
  Interventions: Drug: Tenecteplase
- Alteplase (Active Comparator): Alteplase
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Tenecteplase — 0.4 mg/kg single bolus intravenously
  Other Names: Metalyse
  Arms: Tenecteplase
Drug: Alteplase — 0.9 mg/kg as 10% bolus + 90% infusion/60 minutes intravenously
  Other Names: Actilyse
  Arms: Alteplase

SUMMARY:
Background: Alteplase is the only approved acute drug treatment in ischemic stroke and aims at dissolving arterial clots causing cerebral ischemia. The overall benefit of alteplase is substantial. However, there is considerable room for improvement as 2/3 of patients with large clots may not achieve reopening of the vessel and up to 40% of the patients remain severely disabled or die.

Tenecteplase, a modified tissue plasminogen activator, has been shown to be a more efficient and safer thrombolytic drug than alteplase in pre-clinical studies. Tenecteplase has replaced alteplase as thrombolytic treatment in myocardial infarction and may also be the drug of choice in ischemic stroke.

Tenecteplase and alteplase had a similar safety profile in the NOR-TEST trial and there were no differences in efficacy between the two treatment groups. However, a majority of patients had mild stroke which may be associated with a natural favorable prognosis.

In spite of these neutral results, tenecteplase has the potential to replace alteplase as the drug of choice, based on a better pharmacological profile and a simpler practical administration. There is, however, need for a higher number of patients to prove the efficacy and safety of tenecteplase.

Hypothesis: Tenecteplase 0.4 mg/kg is non-inferior compared with alteplase 0.9 mg/kg.

DETAILED DESCRIPTION:
Objectives: To compare efficacy and safety of tenecteplase 0.4 mg/kg (single bolus) vs. alteplase 0.9 mg/kg (10% bolus + 90% infusion/60 minutes) a) within 4½ hours after symptom onset; b) within 4½ hours after awakening with stroke symptoms, and c) as bridging therapy within 4½ hours before thrombectomy.

Study design: NOR-TEST-2 is a multi-centre PROBE (prospective randomised, open-label, blinded endpoint) trial, designed to establish non-inferiority of tenecteplase as compared with alteplase for consecutively admitted patients with acute ischaemic stroke treated within 4½ hours after symptom onset. Randomisation tenecteplase:alteplase is 1:1.

Endpoints: Primary endpoint is functional outcome (mRS 0-1) at 90 days (efficacy). Secondary endpoints include rates of cerebral hemorrhages on CT/MR at 24-48 hours and mortality (safety).

Patient recruitment: All patients admitted to hospital with acute ischaemic stroke eligible for standard iv thrombolysis with alteplase and with pre-stroke mRS<3 and NIHSS score of >5 on admission are potentially eligible for NOR-TEST-2. Based on power calculations from NOR-TEST, NOR-TEST 2 aims at including 1036 patients.

ELIGIBILITY:
General inclusion criteria

* 18 years or older
* Ischaemic stroke with clinical symptoms corresponding to National Institutes of Health Stroke Scale Score (NIHSS) of >5. All stroke sub-types and vascular distributions are eligible. A visible arterial occlusion is not required for inclusion.
* Treatment <4½ hours after stroke onset or after awakening with symptoms.
* Informed consent by patient or by patient's family

Specific sub-set inclusion criteria

* Wake-Up Stroke: FLAIR-DWI mismatch on MRI as judged by the (neuro-) radiologist or neurologist.
* Thrombectomy: Occlusion of intracerebral artery technically accessible for endovascular embolectomy as defined by local treatment protocols.

Exclusion criteria

* Prestroke modified rankin scale of ≥3
* Large areas of hypodense ischaemic changes on baseline CT;
* Patients with systolic blood pressure >185 mm Hg or diastolic blood pressure >110 mm Hg in spite of acute antihypertensive treatment;
* Pregnant women (are treated with alteplase);
* Women with possible pregnancy (are treated with alteplase)
* Beast feeding women, if a 24 hours stop of feeding is not feasible.
* Clinical presentation suggesting subarachnoid haemorrhage even if baseline CT is normal;
* Known bleeding diathesis; use of oral anticoagulants with no antidot, INR ≥1,4; heparin <48 hours and increased APTT; low molecular weight heparin(oid) <24 hours; another investigational drug <14 days;
* Patients with arterial puncture at a noncompressible site or lumbar puncture <7 days; major surgery or serious trauma <14 days; gastrointestinal or urinary tract hemorrhage <14 days; clinical stroke <2 months; history of intracranial haemorrhage; CNS neurosurgery <2 months; serious head trauma <2 months; pericarditis; sepsis; any serious medical illness likely to interact with treatment; confounding pre-existent neurological or psychiatric disease; unlikely to complete follow-up;
* Any condition that, in the opinion of the investigator, puts a patient at risk if treated with thrombolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with favorable functional outcome | 90 days
  Modified Rankin Scale 0-1 (favorable= 0-1, unfavorable 2-6)

SECONDARY OUTCOMES:
Symptomatic cerebral hemorrhage | 24-48 hours
  Proportion of patients with haemorrhagic infarct/haematoma as defined by CT or MRI
Any cerebral haemorrhage | 24-48 hours
  Proportion of patients haemorrhagic infarct/haematoma as defined by CT or MRI
Major neurological improvement | 24 hours
  Proportion of patients >3 Points improvement by NIHSS score or NIHSS score 0 (NIHSS score range is 0-42)
Functional handicap | 90 days
  Ordinal shift analysis of modified Rankin scale (0-6)
Mortality | 90 days
  Proportion of patients who died

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, Thommessen B, Amthor KF, Ihle-Hansen H, Kurz M, Tobro H, Kaur K, Stankiewicz M, Carlsson M, Morsund A, Idicula T, Aamodt AH, Lund C, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017 Oct;16(10):781-788. doi: 10.1016/S1474-4422(17)30253-3. Epub 2017 Aug 2. PMID 28780236
- [Result] Kvistad CE, Naess H, Helleberg BH, Idicula T, Hagberg G, Nordby LM, Jenssen KN, Tobro H, Rorholt DM, Kaur K, Eltoft A, Evensen K, Haasz J, Singaravel G, Fromm A, Thomassen L. Tenecteplase versus alteplase for the management of acute ischaemic stroke in Norway (NOR-TEST 2, part A): a phase 3, randomised, open-label, blinded endpoint, non-inferiority trial. Lancet Neurol. 2022 Jun;21(6):511-519. doi: 10.1016/S1474-4422(22)00124-7. Epub 2022 May 4. PMID 35525250
- [Derived] Novotny V, Kvistad CE, Naess H, Logallo N, Fromm A, Khanevski AN, Thomassen L. Tenecteplase, 0.4 mg/kg, in Moderate and Severe Acute Ischemic Stroke: A Pooled Analysis of NOR-TEST and NOR-TEST 2A. J Am Heart Assoc. 2023 Oct 17;12(20):e030320. doi: 10.1161/JAHA.123.030320. Epub 2023 Oct 13. PMID 37830342